CLINICAL TRIAL: NCT02019836
Title: Comparison of Maternal and Neonatal Vitamin D Levels in Term Neonates With and Without Early Onset Sepsis
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merih Cetinkaya, Associate Professor, MD, PhD, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: MC10000
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Vitamin D Deficiency
Keywords: vit D; sepsis; newborn; maternal; neonatal
MeSH Terms: conditions — Vitamin D Deficiency; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- sepsis group, control group: Sepsis group; infants with the diagnosis of high probable sepsis Control group; infants without sepsis
  Interventions: Other: Determining maternal and neonatal vitamin D levels

INTERVENTIONS:
Other: Determining maternal and neonatal vitamin D levels

SUMMARY:
Neonatal sepsis is a clinical syndrome characterized by signs and symptoms of infection with or without accompanying bacteremia in the first month of life which is still an important cause of morbidity and mortality. Vitamin D is a fat-soluble steroid hormone that primarily contributes to the maintenance of normal calcium homeostasis and skeletal mineralization. In addition to its classical role in bone metabolism, vitamin D also has immunomodulatory effects on immune function. Although some studies reported a link between vitamin D deficiency and critical illness in adults, a direct relationship has not been directly shown yet. However, to the best of our knowledge, no study evaluated the association between EOS and maternal/neonatal vitamin D levels. The objective of this prospective study is to determine the possible role of maternal and neonatal plasma vitamin D levels on EOS development in term infants. We also aim to evaluate possible effect of the severity of vitamin D deficiency on EOS development in the study population.

DETAILED DESCRIPTION:
Term infants with clinical and laboratory findings of early onset sepsis who are >37 weeks of gestational age and will be admitted to Neonatal Care Unit of Kanuni Sultan Suleyman Training and Research Hospital will be included in this prospective study. The study group will consist of term neonates who are clinically suspected to have an early infection from the 1st day of life. Blood for neonatal and maternal vitamin D levels will be obtained from all infants and their mothers at the time of hospital admission. Only infants with high probable sepsis will consist the study group. The healthy infants who admit to our outpatient clinic for routine evaluation at postnatal day 3 with no signs of clinical and laboratory infection and are evaluated for hyperbilirubinemia will be referred to as the Control group. The Control group wll consist term infants with the same gestational and postnatal age of the infants that will be included in the study group. In both groups, maternal samples will be obtained at the postpartum period at the time of infant's hospitalization. Plasmas after separated and stored at -800C. Levels of 25-OHD were determined using Shimadzu LC-20AT model High Performance Liquid Chromatography (HPLC) system. Data will be analyzed using SPSS software and appropriate statistical analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Infants >37 weeks of gestational age and are admitted to Neonatal Care Unit of Kanuni Sultan Suleyman Training and Research Hospital
* Infants with clinical and laboratory findings of early neonatal sepsis
* Term infants without sepsis as the control group

Exclusion Criteria:

* presence of maternal clinical and/or histological chorioamnionitis,
* presence of premature rupture of membranes (PROM),
* infants with probable or possible sepsis according to criteria,
* refusal of parental consent,
* lack of laboratory data,
* major congenital abnormalities

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants admitted to neonatal care unit with the diagnosis of high probable sepsis will constitute the sepsis group, whereas infants admitted to outpatient clinic without findings of sepsis will constitute the control group
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
development of early onset sepsis | 1 year
  A total of 100 infants will be included and vitamin D levels will be compared between those with and without neonatal sepsis

SECONDARY OUTCOMES:
severity of vitamin D deficiency and neonatal sepsis | one year
  Infants will be divided into three groups in terms of mild, moderate and severe vitamin D deficiency according to maternal and neonatal vitamin D levels and a possible association between vitamin D deficiency and culture proven sepsis will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Merih Cetinkaya, Study Director — Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Gitto E, Karbownik M, Reiter RJ, Tan DX, Cuzzocrea S, Chiurazzi P, Cordaro S, Corona G, Trimarchi G, Barberi I. Effects of melatonin treatment in septic newborns. Pediatr Res. 2001 Dec;50(6):756-60. doi: 10.1203/00006450-200112000-00021. PMID 11726736
- [Background] Karatekin G, Kaya A, Salihoglu O, Balci H, Nuhoglu A. Association of subclinical vitamin D deficiency in newborns with acute lower respiratory infection and their mothers. Eur J Clin Nutr. 2009 Apr;63(4):473-7. doi: 10.1038/sj.ejcn.1602960. Epub 2007 Nov 21. PMID 18030309